CLINICAL TRIAL: NCT03042117
Title: Connecting Periodontal and Coronary Artery Disease Via the Inflammatory State of the Body
Status: Withdrawn | Type: Observational
Why Stopped: Insufficient funds
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Other Study IDs: L17-008
Record Dates: First submitted 2017-01-26; First posted 2017-02-03 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Periodontal Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Periodontal Diseases; Cardiovascular Diseases | interventions — Periodontal Index

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- No Coronary Artery Disease (CAD): Patients with no known cardiovascular disease.
  Interventions: Other: periodontal probing
- CAD without Myocardial Infarction (MI): Patients with cardiovascular disease without a myocardial infarction.
  Interventions: Other: periodontal probing
- CAD with MI: Patients with cardiovascular disease with previous history of a myocardial infarction.
  Interventions: Other: periodontal probing

INTERVENTIONS:
Other: periodontal probing — A periodontal probe will be inserted between the tooth and the gum in the gingival sulcus and a measurement of the pocket depth will be measured by a trained dentist in all subjects

SUMMARY:
Cardiovascular disease is one of the leading causes of death in the United States and the world. Many interventions relating to prevention have been emphasized as more risk factors for this devastating disease are discovered. Periodontal disease is known to have a close association with cardiovascular disease, but its role as a risk factor is still not well understood. Inflammation is a driving force in both of these diseases, creating a potential bridge between the two. Specifically, periodontal disease can cause an inflammatory reaction in the body, which may predispose or even directly contribute to atheroma formation in the coronary arteries. In this study, the investigators will study the link between the inflammatory state of the body and will search for a correlation with levels of coronary artery disease and periodontal disease. Inflammatory markers such as high-sensitivity C-reactive protein (hs-CRP), erythrocyte sedimentation rate (ESR), and immunoglobulin G (IgG) levels in the patient's blood will be analyzed and correlated to clinical attachment loss measured via pocket depth measurement, the distance from the gingival margin to the base of the pocket. A definitive link between these disease processes will allow preventive measures to be taken earlier to prevent this lifelong disease.

DETAILED DESCRIPTION:
Dental probes will be used to probe depth of gum recession in subjects with and without a history of cardiac events. Venous blood samples will also be collected from all subjects for measurement of sedimentation rate, myeloperoxidase, and IgG levels. Statistical analysis will then be done, in attempt to identify a difference in gum recession depth and/or serum inflammatory markers among those with and without prior cardiac events.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with known CAD with previous MI, OR
2. Patients without known CAD
3. Ages 18-89 years
4. Patients who have dental implants with a recorded patient history of how the teeth were lost
5. Patients with at least one tooth in each of the four quadrants of the mouth
6. Able to obtain all necessary pocket measurements and blood samples needed for the study

Exclusion Criteria:

1. Patients with a known history of rheumatoid arthritis
2. Patients with a known history of lupus
3. Patients currently under the care of a rheumatologist
4. Patients who have had a MI in the two weeks prior to entering the study
5. Patients with a previous history of coronary artery bypass graft
6. Current smokers and tobacco users
7. Patients on disease-modifying agents for rheumatoid arthritis (methotrexate)10. Patients who have undergone chemotherapy in the past five years
8. Patients who currently use steroids or immunosuppressive agents

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients from ages 18-89 years who are being seen in the Center for Cardiovascular Health at TTUHSC and at Dr. Johnson's dental clinic who meet the inclusion criteria, and who will consent to participating in the study. There will be between 25 to 35 patients in each group.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
Level of periodontal disease | one day

SECONDARY OUTCOMES:
ESR | one day
Myeloperoxidase (MPO) | one day
IgG | one day
hs-CRP | one day

CONTACTS AND LOCATIONS:
Overall Officials: Ami Knox, MBA, Study Director — Texas Tech University Health Sciences Center

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with other researchers